CLINICAL TRIAL: NCT06935656
Title: Effectiveness of Three Executive Function Interventions on Direct and Far Transfer in Chilean School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, nicholas napolitano, Principal Investigator, University of Talca
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 21231300; 45/2024 (Other: University of Talca Scientific Ethics Committee)
Record Dates: First submitted 2025-04-04; First posted 2025-04-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Executive Functions
Keywords: Executive functions; intervention; academic performance

STUDY DESIGN:
Intervention Model Description: This cluster-randomized, between-subjects factorial study examines two independent variables: (1) intervention modality (digital, traditional, mixed, and control) and (2) age group (5-6, 9-10 years), forming a 4 × 2 design with eight groups. Four schools will be randomly assigned to one modality. All follow the same state curriculum and serve demographically similar urban children, ensuring baseline comparability. Within each school, both age groups will participate, allowing analysis of main and interaction effects. The intervention delivers the same EF program via digital, traditional, or mixed formats, while the control group receives no specialized EF training. Executive functions, literacy, and math will be measured pre- and post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5-6 year old group (Experimental): This arm is made up of the younger group of participants (aged 5-6 years old) who will be randomly assigned to one of the three interventions.
  Interventions: Other: Tablet-based executive function intervention; Other: Traditional executive function intervention; Other: Mixed executive function intervention
- 9-10 year old group (Experimental): This arm is made up of the older group of participants (aged 9-10 years old) who will be randomly assigned to one of the three interventions.
  Interventions: Other: Tablet-based executive function intervention; Other: Traditional executive function intervention; Other: Mixed executive function intervention
- 5-6 year old TAU group (No Intervention): This arm is made up of the younger group of participants (aged 5-6 years old) who will be randomly assigned to no intervention, and will receive their normal schooling.
- 9-10 year old TAU group (No Intervention): This arm is made up of the older group of participants (aged 9-10 years old) who will be randomly assigned to no intervention, and will receive their normal schooling.

INTERVENTIONS:
Other: Tablet-based executive function intervention — This intervention contains activities that have been designed to stimulate the development of children's executive functioning (working memory, inhibitory control and cognitive flexibility). Each activity is presented in a gamified environment, and each executive function is stimulated for an equal amount of time through activities that children complete on a tablet.
  Arms: 5-6 year old group; 9-10 year old group
Other: Traditional executive function intervention — This intervention contains activities that have been designed to stimulate the development of children's executive functioning (working memory, inhibitory control and cognitive flexibility). Each activity is presented as a game, and each executive function is stimulated for an equal amount of time through activities that require motor skills, the manipulation of cards and the use of paper and pencil tasks.
  Arms: 5-6 year old group; 9-10 year old group
Other: Mixed executive function intervention — This intervention contains activities that have been designed to stimulate the development of children's executive functioning (working memory, inhibitory control and cognitive flexibility). Each activity is presented as a game, and each executive function is stimulated for an equal amount of time. Half of the intervention sessions utilize activities that require motor skills, the manipulation of cards and the use of paper and pencil tasks, and the other half are activities that are completed on a tablet.
  Arms: 5-6 year old group; 9-10 year old group

SUMMARY:
Executive functions (EF) are a set of effortful cognitive processes that allow children to control their thoughts, emotions, behaviors, update information in their memory and be mentally flexible. The literature shows that the development of EF is essential for school success, in addition to being an important predictor of quality of life in adulthood. As a result, numerous interventions have sought to stimulate EF development through different programs and formats, typically reporting moderate effectiveness in improving core EF components. However, evidence for effects on untrained, domain-specific areas, such as academic performance, is less consistent. One explanation for these mixed findings may lie in the heterogeneity of interventions and participant characteristics; particularly regarding the modality of the intervention (e.g., using digital media versus traditional media) and children's stage of development. Although the current literature suggests these factors moderate intervention efficacy, there is a lack of randomized controlled trials that compare these variables within a single design. To address this gap, a randomized controlled study has been proposed, aimed at examining an EF intervention delivered in one of three modalities-traditional (paper-and-pencil), digital (computer-based), and mixed-in low-income, urban Chilean school children at two developmental stages (5-6 years and 9-10 years). Each program will target core EF components and measure both efficacy in EF improvement and outcomes in literacy and math skills. By contrasting these intervention modalities across distinct age groups, this study seeks to identify whether developmental level and format have moderating effects on EF improvement and academic performance. Our findings will contribute to ongoing debates about the best practices for EF stimulation, potentially informing evidence-based interventions that can be scaled or adapted for children at different developmental stages and in under-resourced settings. In doing so, this research seeks to clarify how, when, and for whom EF interventions yield lasting benefits beyond immediate cognitive skills.

ELIGIBILITY:
Inclusion Criteria:

* Schools must be classified by the Chilean government as being public elementary schools located in an urban setting, with a proportion of vulnerability of at least 70% or greater (index for socioeconomic status). Schools also must contain at least one kindergarten class.
* For participants, the children must be regularly attending either kindergarten, or the fourth or fifth grade.

Exclusion Criteria:

* Schools that are considered rural, private or subsidized are not eligible. Additionally, schools that have a vulnerability index of less than 70% are not eligible.
* For participants, children with an intellectual disability, or are unable to understand and speak Spanish, will be excluded from the data analysis.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in working memory | From baseline to end of intervention at 12 weeks
  Working memory will be measured using a direct task known as the Corsi Block Test. The test has an internal consistency of 0.93 (95% confidence interval of 0.84 - 0.97) in children ages 10-11 years. Participants will see nine blocks on a screen. The participant will be instructed to watch a sequence of blocks that illuminate. The participant will need to replicate the sequence by touching the blocks on the screen. Sequences begin simple (2 blocks) and become more difficult throughout the trials (up to 9 blocks). A score is determined by the number of errors and the number of correct responses. A higher score indicates better working memory.
Change from baseline in inhibitory control | From baseline to end of intervention at 12 weeks
  To measure inhibitory control, the Hearts and Flowers task will be used. Participants will watch a stimulus of either a heart or a flower in the center of a screen. In the congruent trials, participants will respond with the same stimulus by touching either the smaller heart or flower to the left or right (respectively) of the main stimulus on screen. In the incongruent trials, the opposite of the stimulus must be touched. Reaction time and accuracy are both collected from each trial. Lower reaction time and more accurate responses indicate better inhibitory control. This task was adapted in Chile and had a Cronbach's alpha of 0.83 in children aged 6 to 10 years.
Change from baseline in cognitive flexibility | From baseline to end of intervention at 12 weeks
  Cognitive flexibility will be measured using a modified version of the Dimensional Change Card Sort. This task requires participants to group images on cards first using two dimensions: shape in the first set of trials, then color in the second set. Next, in the third set of trials, participants are asked to group images on cards based on three dimensions: shape, color, or quantity. Reaction time and accuracy are recorded from each trial. Lower reaction time and better accuracy indicate better cognitive flexibility. This instrument has not been validated in Chile but has a reliability coefficient of 0.92 in children aged 6-15 years.

SECONDARY OUTCOMES:
Change from baseline in literacy | From baseline to end of intervention at 12 weeks
  The Tejas LEE instrument will be used to measure literacy. This is a standardized instrument designed for children from kindergarten to third grade. It evaluates various reading competencies through four scales and was adapted in Chile. In each of the scales, higher accuracy of responses indicates better literacy.
Change from baseline in math ability | From baseline to end of intervention at 12 weeks
  The Woodcock-Muñoz III Battery will be used to measure mathematical skills. This test was adapted from English to Spanish and contains several subtests designed to assess mathmatical skills. In each of the subtests, higher accuracy scores indicate better math skills. Among Spanish-speaking children aged four to 13 years, the reliabilities of these subtests range between 0.84 and 0.97.

CONTACTS AND LOCATIONS:
Locations (5):
- Chile (5):
  - Municipal School 2, Talca, Maule Region
  - Municipal School 4, Talca, Maule Region
  - Municipal School 5, Talca, Maule Region
  - Municipal School 1, Talca, Maule Region
  - Municipal School 3, Talca, Maule Region

IPD SHARING:
Plan to Share IPD: Yes
The study will follow open science guidelines in that the anonymized data and the R analysis script will be made available on the OSF registry of this study. Parents and guardians will be informed of this process in the informed consent form.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The protocol, SAP and ICF are currently available on the OSF study registry (start date: March 11, 2025). Analytic code will be when the statistical analyses are complete (estimated date: June, 2026). This data will be available for five years, as per guidelines set by the University of Talca's Scientific Ethics Commitee.
Access Criteria: Anyone with the provided link will be able to access this information.
URL: https://osf.io/9mp83

REFERENCES:
- [Derived] Napolitano N, Rojas-Barahona CA, Gaete J, Araya R. A comparison of three executive function interventions on direct and far transfer in Chilean school children: a cluster-randomized controlled protocol. BMC Psychol. 2025 Jul 4;13(1):730. doi: 10.1186/s40359-025-03075-3. PMID 40615866
- See also: Study protocol — https://osf.io/9mp83
- Available data/document: All of the information regarding the Consent forms, IRB certificate as well as the analytic code and data can be found here.: DOI 10.17605/OSF.IO/Y4SGJ — https://osf.io/y4sgj/files/osfstorage/67d6ddfb6a60610ab9a72a9b — The analytic code and data will be uploaded once the data is collected (est. December, 2025) and analyzed (est. June, 2026)
- Available data/document: Study Protocol — https://osf.io/9mp83